CLINICAL TRIAL: NCT03796234
Title: Multidisciplinary Program Based in High Intensity Interval Training and Dietary Education for Coronary Artery Disease With Percutaneous Coronary Intervention
Brief Title: Multidisciplinary Program Based in High Intensity Interval Training and Dietary Education for Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, Doctor in Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 147697976792
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Diet; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary and physiotherapy (Experimental): A multidisciplinary program was developed. 3 group talks were carried out, in a period of 3 months, in which different topics related to healthy eating were treated. In addition, a 3-month high intensity interval training program was developed. Physiotherapy sessions were carried out twice a week for one hour and intensity was established based in effort tests.
  Interventions: Other: Dietary and physiotherapy
- Physiotherapy (Experimental): A 3-month high intensity interval training program was developed. Physiotherapy sessions were carried out twice a week for one hour and intensity was established based in effort tests.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Dietary and physiotherapy — 3 group talks were carried out, in a period of 3 months, in which different topics related to healthy eating were treated. In addition, a 3-month high intensity interval training program was developed. Physiotherapy sessions were carried out twice a week for one hour and intensity was established based in effort tests.
  Arms: Dietary and physiotherapy
Other: Physiotherapy — A 3-month high intensity interval training program was developed. Physiotherapy sessions were carried out twice a week for one hour and intensity was established based in effort tests.
  Arms: Physiotherapy

SUMMARY:
A multidisciplinary program based on physiotherapy and diet education will be carried out for 3 months in patients with coronary artery disease with percutaneous coronary intervention. Educational lectures on nutrition and high intensity interval training will be developed in old patients with chronic heart disease. A control group will not develop any program. Effectiveness on anthropometric parameters, eating habits, physical activity, quality of life, anxiety and depression will be assessed at baseline and at 3 months.

DETAILED DESCRIPTION:
A multidisciplinary program based on high intensity interval training and diet education will be carried out for 3 months for patients with coronary artery disease with percutaneous coronary intervention. Three educational lectures on nutrition and a 3-month high intensity interval training will be developed in old patients with chronic heart disease. A control group will not develop any program. Effectiveness on anthropometric parameters, eating habits, physical activity, quality of life, anxiety and depression will be assessed at baseline and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* infarction or angina pectoris.
* At least six months elapsed since the diagnosis of heart disease at the time of the start of the study.
* Be physically and cognitively able to complete the evaluations and the program.

Exclusion Criteria:

* Present another type of cardiac disease different from ischemic heart disease.
* Present any physical or psychiatric condition that prevents the normal performance of the evaluations and the program.
* Mobility problems to attend reassessments.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Adherence to the mediterranean diet | baseline
  Test of adherence to the mediterranean diet, which consists of 14 questions related to the Mediterranean diet. Depending on the answer of the question it can be obtained 1 point or 0 points, being the value of each item 0 or 1. If the sum of the points is 9 or higher the subject has a good adhesion to the mediterranean diet. If it is less than 9 points is considered bad adhesion. The range can vary between 0 points (minimum adhesion) and 14 points (maximum adhesion) (PREDIMED, 2017).
Adherence to the mediterranean diet | 3 months
  Test of adherence to the mediterranean diet, which consists of 14 questions related to the Mediterranean diet. Depending on the answer of the question it can be obtained 1 point or 0 points, being the value of each item 0 or 1. If the sum of the points is 9 or higher the subject has a good adhesion to the mediterranean diet. If it is less than 9 points is considered bad adhesion. The range can vary between 0 points (minimum adhesion) and 14 points (maximum adhesion) (PREDIMED, 2017).
Food consumption frequency questonnaire | baseline
  Food consumption frequency questionnaire: registers the number of times/week or the number of times/month a series of foods is consumed, so that information about the foods the individual consumes most frequently during the week can be obtained. The list of foods that are part of the questionnaire is made up of those most common among the population, with a total of 45 items (yoghurts, fish, fruits, etc.). It also includes a table called Table of Weight of the Item Ration (PRI), in which the weight of the ration of each item is collected to facilitate the completion of the questionnaire (Trinidad et al., 2008).
Food consumption frequency questonnaire | 3 months
  Food consumption frequency questionnaire: registers the number of times/week or the number of times/month a series of foods is consumed, so that information about the foods the individual consumes most frequently during the week can be obtained. The list of foods that are part of the questionnaire is made up of those most common among the population, with a total of 45 items (yoghurts, fish, fruits, etc.). It also includes a table called Table of Weight of the Item Ration (PRI), in which the weight of the ration of each item is collected to facilitate the completion of the questionnaire (Trinidad et al., 2008).

SECONDARY OUTCOMES:
Body composition: body fat in %, visceral fat in %, muscle mass in %, body water in % | baseline
  Bioimpedanciometer OMRON HBF-500INT
Body composition: body fat in %, visceral fat in %, muscle mass in %, body water in % | 3 months
  Bioimpedanciometer OMRON HBF-500INT
Weight (in kilograms) | baseline
  Weight (in kilograms)
Weight (in kilograms) | 3 months
  Weight (in kilograms)
Body mass index | baseline
  weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2
Body mass index | 3 months
  weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2
Circumferences: abdominal circumference in cm, hip circumference in cm, arm circumference in cm, calf circumference in cm | baseline
  Circumferences by using a measuring tape
Circumferences: abdominal circumference in cm, hip circumference in cm, arm circumference in cm, calf circumference in cm | 3 months
  Circumferences by using a measuring tape
Triceps fat fold in mm | Baseline
  Lipocalibre Holtain
Triceps fat fold in mm | 3 months
  Lipocalibre Holtain
Physical activity | baseline
  International physical activity questionnaire: it has 9 items and provides information on the time spent while walking, in activities of low, moderate and vigorous intensity and in sedentary activities. Based on the estimated METS consumed, the IPAQ divides the subjects into three levels or categories: Low, moderate and high physical activity.
  The score of the different types of activity is expressed in METS-minutes per week.
Physical activity | 3 months
  International physical activity questionnaire: it has 9 items and provides information on the time spent while walking, in activities of low, moderate and vigorous intensity and in sedentary activities. Based on the estimated METS consumed, the IPAQ divides the subjects into three levels or categories: Low, moderate and high physical activity.
  The score of the different types of activity is expressed in METS-minutes per week.
Health related quality of life | baseline
  Short-form 36: the questionnaire is composed of 36 questions that value both positive and negative health status. It was developed from an extensive battery of questionnaires employed at WHO, which included 40 concepts related to health. The questionnaire contains 8 scales, which represent the concepts of health most frequently used in the main health questionnaires. The 36 items of the instrument cover the following scales: Physical function, Physical role, Body pain, General health, Vitality, Social function, Emotional role, Mental health. The scores of each of the 8 dimensions of the SF-36 oscillate between 0 and 100. A result of 100 indicates optimal health and 0 would reflect a very poor state of health.
Health related quality of life | 3 months
  Short-form 36: the questionnaire is composed of 36 questions that value both positive and negative health status. It was developed from an extensive battery of questionnaires employed at WHO, which included 40 concepts related to health. The questionnaire contains 8 scales, which represent the concepts of health most frequently used in the main health questionnaires. The 36 items of the instrument cover the following scales: Physical function, Physical role, Body pain, General health, Vitality, Social function, Emotional role, Mental health. The scores of each of the 8 dimensions of the SF-36 oscillate between 0 and 100. A result of 100 indicates optimal health and 0 would reflect a very poor state of health.
Anxiety | baseline
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
Anxiety | 3 months
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
Depression | baseline
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).
Depression | 3 months
  Hospital anxiety and depression questionnaire: the questionnaire includes 14 questions regarding the depressant and anxious symptoms of the patient. Two subsets of 7 items each, on Likert scale 0-3. For anxiety HAD-A sum of odd items (1,3,5,7,9,11,13), for depression HAD-D sum of even items (2,4,6,8,10,12,14 ), with a score range in each subscale of 0-21. A higher score means greater anxiety and depression. For both subscales, scores higher than eleven would indicate "case" and greater than eight would be considered "probable case". The internal consistency for the Spanish population is HAD-A α = .83 and HAD-D α = .87 (Vallejo, Rivera, Esteve-Vives and RodríguezMuñoz, 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Marques-Sule, PT, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No